CLINICAL TRIAL: NCT06706037
Title: Do Reformer Pilates Exercises Change Pain Perception in Patients With Chronic Musculoskeletal Pain?A Comparative Study.
Brief Title: Effect of Reformer Exercises on Pain Perception in Chronic Musculoskeletal Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atılım University (Other)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, Assistant Professor, Atılım University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Atılım2
Record Dates: First submitted 2024-10-08; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Musculoskeletal Pain
Keywords: chronic pain; musculoskeletal pain; reformer pilates
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: prospective cross-sectional randomized controlled study
Who Masked: Participant
Masking Description: The study participants were made to exercise for 6 weeks, but they were not informed about the purpose of the study and evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reformer exercise grup (Experimental): Reformer exercise group will receive a 6-week reformer pilates exercise.
  Interventions: Other: Exercise
- control group (No Intervention): The control group will consist of patients with chronic musculoskeletal pain waiting in the treatment list. No intervention method will be applied to the patients in the control group.

INTERVENTIONS:
Other: Exercise — A 6 week reformer pilates exercise program
  Arms: reformer exercise grup

SUMMARY:
This study was planned to investigate whether reformer pilates exercises, which are recommended for the development and maintenance of well-being in musculoskeletal problems associated with low back, neck and back pain, change the pain perceptions of patients with chronic musculoskeletal diseases by improving the mind-body relationship.

DETAILED DESCRIPTION:
Although many symptoms are observed in musculoskeletal system disorders, pain which progresses gradually and even progresses to the point of causing incapacity for work is the most common. Although musculoskeletal system disorders indicate a very broad concept, it is also observed that low back, neck and back pain are in the first rank in studies conducted worldwide and in our country .Pilates training plays an important role in regaining and maintaining muscle strength, flexibility, endurance and functioning of proprioceptive mechanisms. Although there are many physical activity programmes, Pilates has become an increasingly widespread and recommended physical exercise method worldwide in recent years. The Pilates method is an exercise concept established by Joseph H Pilates in the early 1900s and currently applied to both sick and healthy individuals. Exercises can be performed on a mat and special equipment such as Cadillac, Reformer and Wundachair are also used. Pilates training plays an important role in regaining and maintaining muscle strength, flexibility, endurance and functioning of proprioceptive mechanisms. Therefore, although Pilates exercises are not designed to reduce body weight, they are a good option for sedentary, overweight and obese people who have difficulty in performing traditional exercises .

This study was planned to investigate whether reformer pilates exercises, which are recommended for the development and maintenance of well-being in musculoskeletal problems associated with low back, neck and back pain, change the pain perceptions of patients with chronic musculoskeletal diseases by improving the mind-body relationship.

ELIGIBILITY:
Inclusion Criteria:

Sedantry male and female aged 30-50 years chronic musculoskeletal pain diagnosed for at least 6 months

Exclusion Criteria:

neurological disorders communication and psychiatric disorders

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measurement by Brief Pain Inventory | Up to one month
  Brief Pain Inventory: The questionnaire was developed by Cleeland and Ryan in 1994 . The pain intensity section of the BPI consists of four items that are scored from 0 (no pain) to 10 (worst possible pain), whereas the functional interference section consists of seven items that are scored from 0 (no interference) to 10 (complete interference). A pain severity score is calculated from the mean of the four pain intensity items, and a pain interference score is calculated from the mean of the seven pain interference items
Pain coping assessment by Pain Coping Inventory. | Up to one month
  Pain Coping Scale: The Pain Coping Questionnaire (PCQ) is a 39-item self-report measure for evaluating pain coping in children and adolescents in both clinical and research settings.16 It consists of 8 subscales that can be categorized into 3 higher-order factors, including approach (composed of information seeking, problem-solving, and seeking social support subscales), problem-focused avoidance (composed of positive self-statements, behavioural distraction, and cognitive distraction subscales), and emotion-focused avoidance (composed of externalizing and internalizing/catastrophizing subscales).
Pain beliefs assessment by Pain Beliefs Scale. | 1month
  Pain Beliefs Scale: It was developed to evaluate the beliefs about the cause and treatment of pain in individuals with pain complaints.Pain beliefs and perceptions inventory (PBAPI).
  The PBAPI was made up to 16 items selected from the piloted version of the PBAPI. Twelve of the items were selected to represent the factors found in the pilot study. Four additional items from the piloted version were included which demonstrated good internal consistency when piloted and which measured the degree to which pain is believed to be a mysterious experience. Each item was presented along with a 4-point Likert scale anchored at the hash marks with degrees of agreement or disagreement.

SECONDARY OUTCOMES:
Kinesiophobia assessment by Tampa Kinesiophobia Scale | 1 month
  Tampa Kinesiophobia Scale: The Tampa Kinesiophobia Scale measures fear of movement/reinjury.Individual item scores range from 1-4, with the negatively worded items (4,8,12,16) having a reverse scoring (4-1). The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Fatigue assessment by Functional Assessment of Chronic Illness Therapy. | 1 month
  FACIT Fatigue The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued).Score range is 0-52.Less than 30 score shows severe fatique.
Sleep quality assessment | 1 month
  Pittsburg Sleep Quality Index: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Şahan, Principal Investigator — Çankırı KaratekinvUniversity, Ankara/TURKEY
Locations (1):
- Naime Ulug, Ankara, Select State, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahan N, Ulug N, Ozeren A. Effects of reformer pilates on pain, psychological factors, and sleep in chronic musculoskeletal pain: a randomized controlled trial. BMC Psychol. 2025 Jul 26;13(1):836. doi: 10.1186/s40359-025-03207-9. PMID 40713915